CLINICAL TRIAL: NCT03602339
Title: LowEr Administered Dose With highEr Relaxivity: Gadovist vs Dotarem (LEADER 75)
Brief Title: Comparison of Gadovist 75% Standard Dose to Dotarem at Full Standard Dose
Acronym: LEADER 75
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 19773; 2018-000690-78 (EudraCT Number)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Magnetic Resonance Imaging
Keywords: Gadolinium; Contrast enhancement; Central nervous system lesion
MeSH Terms: interventions — gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; gadoterate meglumine; ferumoxtran-10; gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1_Suspected CNS-lesion (Experimental): Patients with suspected or confirmed CNS-lesions underwent unenhanced MRI, and contrast-enhanced MRI after gadoterate injection.
  Interventions: Drug: Gadoterate (Dotarem/Clariscan)
- Arm 2_Confirmed CNS-lesion (Experimental): Patients with gadoterate-confirmed CNS-lesions (subgroup of Arm 1) underwent a second unenhanced MRI, and contrast-enhanced MRI after gadobutrol injection.
  Interventions: Drug: Gadoterate (Dotarem/Clariscan); Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadoterate (Dotarem/Clariscan) — Patients received a single dose of 0.5 molar gadoterate (0.1 mmol per kg body weight) intravenously.
  Other Names: Gadoterate
Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875) — Patients received a single dose of 1.0 molar BAY86-4875 (0.075 mmol per kg body weight) intravenously.
  Other Names: Gadobutrol
  Arms: Arm 2_Confirmed CNS-lesion

SUMMARY:
The study was conducted to gain knowledge about a new dose of a diagnostic drug that is used for contrast-enhanced Magnetic Resonance Imaging (MRI) of the human central nervous system (CNS). MRI can visualize the anatomy of the body and is used to detect medical conditions. Diagnostic drugs like gadobutrol and gadoterate contain an element called gadolinium that is applied to improve the analysability of MRI-images.

The purpose of this study was to examine if contrast-enhanced MRI using a reduced dose of the gadolinium-based contrast agent gadobutrol delivers images of similar quality to those obtained when a full dose of the gadolinium-based contrast agent gadoterate was used.

DETAILED DESCRIPTION:
The study was an open-label, multi-center, comparative, cross-over trial in adult patients with known or highly suspected CNS pathology who were referred for imaging of the CNS.

The primary objective of the study was to demonstrate the non-inferiority of gadobutrol (0.075 mmol/ kg body weight) to gadoterate (0.1 mmol/ kg body weight).

ELIGIBILITY:
Inclusion Criteria:

* Known or highly suspected central nervous system (CNS) pathology referred for contrast-enhanced MRI of the CNS.
* Glomerular filtration rate (eGFR) value ≥ 60 mL/min/1.73m2 derived from a serum creatinine result within four weeks prior to the first study MRI.
* Women with negative urine pregnancy test within 1 hour prior to the administration of gadoterate (the first MRI).

Exclusion Criteria:

* No enhancing lesion visible on the gadoterate-enhanced MRI scan.
* Pregnancy or breastfeeding.
* Severe cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Mount Sinai Hospital, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- France (2):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU STRASBOURG - Hôpital de Hautepierre, Strasbourg
- Germany (6):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universität Rostock - Medizinische Fakultät, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Leipzig AöR, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein (UKSH), Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein / AÖR, Lübeck, Schleswig-Holstein
  - Friedrich-Schiller-Uni. Jena, Jena, Thuringia
- Italy (3):
  - ASL Provincia di Barletta-Andria-Trani, Andria, Apulia
  - A.O.U. Pisana, Pisa, Tuscany
  - ULSS2 Marca Trevigiana, Treviso, Veneto
- South Korea (2):
  - Ulsan University Hospital, Ulsan, Ulsan Gwang''yeogsi
  - Seoul National University Hospital, Seoul
- Switzerland (2):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Inselspital Universitätsspital Bern, Bern
- Royal Preston Hospital, Preston, Lancashire, United Kingdom

REFERENCES:
- [Derived] Liu BP, Rosenberg M, Saverio P, Weon YC, Peters S, Ardellier FD, Boeckenhoff A, Endrikat J. Clinical Efficacy of Reduced-Dose Gadobutrol Versus Standard-Dose Gadoterate for Contrast-Enhanced MRI of the CNS: An International Multicenter Prospective Crossover Trial (LEADER-75). AJR Am J Roentgenol. 2021 Nov;217(5):1195-1205. doi: 10.2214/AJR.21.25924. Epub 2021 Jun 16. PMID 34133205
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 7 countries between 14 November 2018 (first participant first visit) and 13 March 2020 (last participant last visit).
Pre-assignment Details: From 166 participants screened, 9 participants were screening failure and a total of 157 participants were enrolled, 157 received study drug for period 1 however 142 received study drug for period 2.
Groups:
- Gadoterate 0.1 mmol/kg BW-Gadobutrol 0.075 mmol/kg BW: Participants received gadoterate at the standard dose of 0.1 mmol/kg body weight (BW) by single intravenous (IV) injection in Study Period 1 and gadobutrol at a dose of 0.075 mmol/kg BW by single IV injection in Study Period 2.
Period: Overall Study
Arm/Group | Gadoterate 0.1 mmol/kg BW-Gadobutrol 0.075 mmol/kg BW
Started (Started period 1 (Gadoterate)) | 157
Completed Period 1 (Gadoterate) | 155
Started Period 2 (Gadobutrol) | 142
Completed (Completed period 2 (Gadobutrol)) | 142
Not Completed | 15
Not completed — Withdrawal by Subject | 9
Not completed — Physician Decision | 2
Not completed — Other reason | 4

BASELINE CHARACTERISTICS:
Arm/Group | Gadoterate 0.1 mmol/kg BW-Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.3) [lower limit 13.3]
Age, Customized [Number; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 0
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 94
  From 65-84 years | 62
  85 years and over | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 109
  More than one race | 0
  Unknown or Not Reported | 19

OUTCOME MEASURES:

1. Primary Outcome: Degree of Lesion Contrast Enhancement
Description: Degree of lesion contrast enhancement is assessed by 3 blinded Readers (Full Analysis Set). Results are presented as the Average Reader score. Blinded Readers scored up to 5 lesions using image sequences and a 4-point scale (1 - No = Lesion not enhanced; 2 - Moderate = Lesion weakly enhanced; 3 - Good = Lesion clearly enhanced; 4 - Excellent = Lesion clearly and brightly enhanced).
Time Frame: Up to 20 days
Population: Full analysis set (FAS) was used for analysis, which is defined as All participants for whom electronic case report form (eCRF) entries and images are available for unenhanced MRI, combined unenhanced and gadobutrol enhanced MRI, and combined unenhanced and gadoterate enhanced MRI.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Gadoterate 0.1 mmol/kg BW: Participants received gadoterate at the standard dose of 0.1 mmol/kg body weight by single intravenous (IV) injection.
- Gadobutrol 0.075 mmol/kg BW: Participants received gadobutrol at a dose of 0.075 mmol/kg body weight by single intravenous (IV) injection.
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale
  Unenhanced | 0.884 (0.252) | 0.863 (0.201)
  Combined unenhanced/enhanced | 3.007 (0.813) | 2.979 (0.837)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (gadobutrol minus unenhanced) - (gadoterate minus unenhanced); Test type: Non-Inferiority — The score to evaluate the non-inferiority is calculated for each subject as (combined unenhanced/gadobutrol-enhanced - unenhanced) - 0.8*(combined unenhanced/gadoterate-enhanced - unenhanced). The 95% CI is based on a t-distribution. The non-inferiority for gadobutrol is achieved if the one-sided p-value for "H0: (gadobutrol minus unenhanced) - 0.8*(gadoterate minus unenhanced) ≤ 0" is lower than 0.025; p < 0.0001, Paired t-test — No type I error adjustment for multiple comparisons is needed because tests on all 3 primary efficacy variables must be significant to demonstrate primary efficacy; Mean Difference (Final Values) = 0.455, 95% CI 2-sided [0.347 to 0.562]

2. Primary Outcome: Lesion Border Delineation
Description: Lesion border delineation is assessed by 3 blinded Readers (Full Analysis Set). Results are presented as the Average Reader score. Blinded readers scored the delineation of up to 5 lesions using image sequences and a 4-point scale (1 - None = No or unclear delineation; 2 - Moderate = Partial delineation; 3 - Good = Almost clear, but incomplete delineation; 4 - Excellent = Clear and complete delineation).
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale
  Unenhanced | 2.279 (0.820) | 2.278 (0.864)
  Combined unenhanced/enhanced | 3.096 (0.781) | 3.099 (0.828)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (gadobutrol minus unenhanced) - (gadoterate minus unenhanced); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0151, Paired t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.180, 95% CI 2-sided [0.017 to 0.342]

3. Primary Outcome: Lesion Internal Morphology
Description: Lesion internal morphology is assessed by 3 blinded Readers (Full Analysis Set). Results are presented as the Average Reader score. Blinded Readers scored the structure and internal morphology of up to 5 lesions using image sequences and a 3-point scale (1 - Poor = Poor visibility; 2 - Moderate = Partial visibility; 3 - Good = Sufficient visibility)
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale
  Unenhanced | 1.835 (0.620) | 1.823 (0.589)
  Combined unenhanced/enhanced | 2.503 (0.496) | 2.484 (0.545)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (gadobutrol minus unenhanced) - (gadoterate minus unenhanced); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0100, Paired t-test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI 2-sided [0.024 to 0.275]

4. Secondary Outcome: Number of Lesions Identified
Description: Number of lesions identified (up to 10) detected by 3 blinded Readers. The mean (SD) number lesions in the Average Reader for gadobutrol and gadoterate in the Full Analysis Set was reported below.
Time Frame: Up to 20 days
Population: Full analysis set (FAS) was used for analysis, which is defined as All subjects for whom electronic case report form (eCRF) entries and images are available for unenhanced MRI, combined unenhanced and gadobutrol enhanced MRI, and combined unenhanced and gadoterate enhanced MRI.
Measure: Mean (Standard Deviation); unit: Number of lesions identified
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Number of lesions identified | 2.064 (2.254) | 2.137 (2.327)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (Gadobutrol - Gadoterate); Test type: Non-Inferiority — Non-inferiority margin is 0.35. If the lower limit of the 95% CI is > -0.35, then non-inferiority is achieved; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [-0.030 to 0.176]

5. Secondary Outcome: Detection of Malignant Disease
Description: The 3 Blinded Readers had to evaluate if the diagnosis resulting from the combined images was malignant disease or not. Each blinded Reader provided a malignant yes/no response. This was compared to the final diagnosis provided by the Investigator. The majority of Readers (2 or 3 Readers agree) was used to calculate sensitivity, specificity, and accuracy - eg. Final Diagnosis - Malignant (Reader 1-yes, Reader 2-no, Reader 3-yes --- Majority Reader yes) - this would be a match for sensitivity.
  The percentage of sensitivity, specificity, and accuracy of detection of malignant disease detected by 3 blinded Readers, gadobutrol versus gadoterate (Full Analysis Set) is reported below for Majority Readers.
Time Frame: Up to 20 days
Population: as for outcome 4
Measure: Number; unit: Percentage (%)
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Percentage (%)
  Accuracy | 70.2 | 70.2
  Sensitivity | 58.7 | 58.7
  Specificity | 91.8 | 91.8
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Accuracy Difference (Gadobutrol - Gadoterate); Test type: Non-Inferiority — Non-inferiority margin = 10%, if the lower limit of the confidence interval > -10%, then non-inferiority is achieved; Difference (Gadobutrol - Gadoterate) = 0.0, 95% CI 2-sided [-3.40 to 3.40] — The 95% confidence intervals are based on McNemar's test
Statistical Analysis 2: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Sensitivity Difference (Gadobutrol - Gadoterate); Test type: Non-Inferiority — Non-inferiority margin = 10%, if the lower limit of the confidence interval > -10%, then non-inferiority is achieved; Difference (Gadobutrol - Gadoterate) = 0.0, 95% CI 2-sided [-5.22 to 5.22] — The 95% confidence intervals are based on McNemar's test
Statistical Analysis 3: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Specificity Difference (Gadobutrol - Gadoterate); Test type: Non-Inferiority — Non-inferiority margin = 10%, if the lower limit of the confidence interval > -10%, then non-inferiority is achieved; Difference (Gadobutrol - Gadoterate) = 0.00, 95% CI 2-sided [0.00 to 0.00] — The 95% confidence intervals are based on McNemar's test. No continuity correction for calculation of the confidence interval was included. Zero cells lead to degenerated confidence interval

6. Secondary Outcome: Confidence in Diagnosis
Description: Diagnostic confidence detected by 3 blinded Readers, gadobutrol vs gadoterate (Full Analysis Set). Blinded Readers rated their confidence in diagnosis according to a 4-point scale (1 - Not confident; 2 - Somewhat confident; 3 - Confident; 4 - Very confident). Results for the Average Reader are reported below.
Time Frame: Up to 20 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale | 3.272 (0.567) | 3.348 (0.591)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (Gadobutrol - Gadoterate); Test type: Other; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [0.011 to 0.140]

7. Secondary Outcome: Image Quality
Description: Comparison of image quality between gadobutrol and gadoterate detected by 3 blinded Readers (Full Analysis Set). Blinded Readers assessed the image quality of gadobutrol- and gadoterate-enhanced images (randomly assigned as left [L] and right [R] image positions) according to a 5-point scale (1- Image R is worse; 2 - Image R is slightly worse; 3- Image R is similar; 4 - Image R is slightly better; 5 - Image R is better). After unblinding of data, the above codes were translated into the following scale: -2 = Gadobutrol image set is worse ; -1 = Gadobutrol image set is slightly worse ; 0 = Image sets are the same ; 1 = Gadobutrol image set is slightly better; 2 = Gadobutrol image set is better. Results for the Average Reader are reported below.
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW-Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141
Scores on a scale | 0.00 (0.61)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW-Gadobutrol 0.075 mmol/kg BW; Comparison of image quality between gadobutrol and gadoterate; Test type: Other; p = 0.9149, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.10 to 0.11]

8. Secondary Outcome: Contrast Enhancement Utilizing an Exploratory Overall Contrast Enhancement Estimation Algorithm
Description: Comparison of contrast enhancement utilizing an overall contrast enhancement estimation algorithm (Full Analysis Set). The exploratory algorithm analyzed the overall enhancement by comparing the axial T1w (longitudinal relaxation time-weighted) enhanced images to the T1w unenhanced images.
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 88 | 89
Scores on a scale
  Relative score | 0.19894 (0.09905) | 0.18564 (0.09028)
  Full image score | 0.05604 (0.08581) | 0.05573 (0.08036)
  Dice score | 0.92984 (0.04293) | 0.92991 (0.05216)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (Gadobutrol-Gadoterate) for Relative score; Test type: Other; Mean Difference (Final Values) = -0.01968, 95% CI 2-sided [-0.03491 to -0.00445]
Statistical Analysis 2: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (Gadobutrol-Gadoterate) for Full image score; Test type: Other; Mean Difference (Final Values) = 0.00586, 95% CI 2-sided [-0.00589 to 0.01762]
Statistical Analysis 3: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Difference (Gadobutrol-Gadoterate) for Dice score; Test type: Other; Mean Difference (Final Values) = 0.00139, 95% CI 2-sided [-0.00471 to 0.00749]

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Number of subjects with treatment-emergent adverse events (TEAEs) (Safety Analysis Set). TEAEs are defined as any AEs that increase in intensity or that are newly developed during the TE period for Study Period 1 or Study Period 2, where TE period for Study Period 1 goes from the first study drug administration in Study Period 1 to 24 hours post-injection, and TE period for Study Period 2 from the first study drug administration in Study Period 2 to 24 hours post-injection.
Time Frame: From the first study drug administration up to 24 hours post injection
Population: The Safety analysis set (SAF) included all enrolled participants who received at least 1 study treatment administration.
Measure: Number; unit: Participants
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 156 | 143
Participants
  Any TEAE | 4 | 1
  Any study drug-related TEAE | 2 | 1
  Any TEAE related to the protocol | 0 | 0
  Any TEAE leading to discontinuation | 0 | 0
  Any TESAE | 0 | 0
  TEAE with outcome death | 0 | 0

10. Post Hoc Outcome: Comparison of Degree of Lesion Contrast Enhancement Detected by Blinded Readers for Combined Image Sets - Equivalence Test
Description: Comparison of degree of lesion contrast enhancement detected by blinded Readers for combined image sets - Equivalence Test (Full Analysis Set). Results are presented as the Average Reader score.
  Blinded Readers scored up to 5 lesions using image sequences and a 4-point scale (1 - No = Lesion not enhanced; 2 - Moderate = Lesion weakly enhanced; 3 - Good = Lesion clearly enhanced; 4 - Excellent = Lesion clearly and brightly enhanced).
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale | 3.007 (0.813) | 2.979 (0.837)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Test type: Equivalence — An equivalence test was calculated using the two one-sided t-tests (TOST) procedure with null hypotheses H01: (gadobutrol - gadoterate) ≤ -0.05 * (gadoterate), and H02: (gadobutrol - gadoterate) ≥ +0.05 * (gadoterate); p = 0.0049, Two one-sided t-tests (TOST) — The overall p-value was calculated as max(p1, p2) where p1 and p2 are the results of null hypotheses H01 and H02 respectively

11. Post Hoc Outcome: Comparison of Border Delineation Detected by Blinded Readers for Combined Image Sets - Equivalence Test
Description: Comparison of border delineation detected by blinded Readers for combined image sets - Equivalence Test (Full Analysis Set). Results are presented as the Average Reader score. Blinded Readers scored the delineation of up to 5 lesions using image sequences and a 4-point scale (1 - None = No or unclear delineation; 2 - Moderate = Partial delineation; 3 - Good = Almost clear, but incomplete delineation; 4 - Excellent = Clear and complete delineation).
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale | 3.096 (0.781) | 3.099 (0.828)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Test type: Equivalence — An equivalence test was calculated using the two one-sided t-tests (TOST) procedure with null hypotheses H01: (gadobutrol - gadoterate) ≤ -0.05 * (gadoterate) and H02: (gadobutrol - gadoterate) ≥ +0.05 * (gadoterate); p = 0.0013, Two one-sided t-tests (TOST) — [p-value comment as in outcome 10, analysis 1]

12. Post Hoc Outcome: Comparison of Internal Morphology Detected by Blinded Readers for Combined Image Sets - Equivalence Test
Description: Comparison of internal morphology detected by blinded Readers for combined image sets - Equivalence Test (Full Analysis Set). Results are presented as the average Reader score. Blinded Readers scored the structure and internal morphology of up to 5 lesions using image sequences and a 3-point scale (1 - Poor = Poor visibility; 2 - Moderate = Partial visibility; 3 - Good = Sufficient visibility).
Time Frame: Up to 20 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Gadoterate 0.1 mmol/kg BW | Gadobutrol 0.075 mmol/kg BW
Number analyzed (Participants) | 141 | 141
Scores on a scale | 2.503 (0.496) | 2.484 (0.545)
Statistical Analysis 1: Comparison: Gadoterate 0.1 mmol/kg BW vs Gadobutrol 0.075 mmol/kg BW; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p = 0.0065, Two one-sided t-tests (TOST) — [p-value comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first study drug administration up to 24 hours post injection
Description: At study start 1 out of 157 participants received gadobutrol instead of gadoterate in study period 1. This participant dropped out and didn't receive gadoterate dose. That's why only 156 out of 157 participants received gadoterate. 156 participants received gadoterate and 143 participants received gadobutrol. 142 participants received both doses - of the 142 - 1 participant's dose extravasated and could not be adequately imaged and was removed from the efficacy population.
Arm/Group | Gadobutrol 0.075 mmol/kg BW | Gadoterate 0.1 mmol/kg BW
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/156
Other Adverse Events (participants affected / at risk) | 1/143 | 4/156
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.075 mmol/kg BW (N=143) | Gadoterate 0.1 mmol/kg BW (N=156)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT03602339/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT03602339/SAP_004.pdf